**TITLE** 

A randomized trial of vaginal prep solutions to reduce bacteria colony counts in patients having a

vaginal surgery.

**INVESTIGATORS** 

Geoffrey Towers, MD, Rose Maxwell, PhD, James Saelens, MD

SUMMARY OR ABSTRACT

This is a randomized trial comparing the effectiveness of 4 vaginal prep solutions

(betadine, baby shampoo, TechniCare and Peridex) on reducing bacterial colony counts during

surgery preparation. Women undergoing a vaginal surgery will be enrolled into the trial prior to

surgery. Target sample size per group is 15 patients. During standard surgical prep, a vaginal

swab will be taken to assess the initial colony counts for aerobic and anaerobic bacteria. After

the initial swab, the vagina will be prepared using one of the prep 4 solutions (betadine, baby

shampoo, TechniCare or Peridex). After a predefined 10 minutes, the area will be re-swabbed to

determine pre-procedure colony counts. A third swab will be taken following completion of the

procedure to determine post-procedure colony counts. Laboratory analyses for raw colony

counts, sensitivities, identification (using MALDI-TOF) will be performed. We expect that there

will be reduced colony counts at the pre-procedure point with baby shampoo having the least

reduction, followed by betadine and TechniCare, then Peridex. Patient reported outcomes for

vaginal itching and burning as well as patient report of any treatment for vaginal infection will be

collected by telephone at 2 days, 2 weeks and 1 month post-surgery.

BACKGROUND AND LITERATURE REVIEW

Antiseptic preparation for surgical incision sites has greatly reduced postoperative infections.

However, surgical site infections (SSI) are still the leading cause of hospitalizations after

Version: 6

surgery. With the application of antiseptic preparation, a reduction in bacterial counts follows.

The rate at which the bacterial counts rise between preparation and incision may be of variation

depending on the surgical antiseptic scrub.

Betadine (Povidone- iodine), Peridex (Chlorhexidine), baby shampoo and TechniCare

(chloroxynel) are all surgical scrubs approved for the preparation of vaginal access surgeries.

While there has been controversy on the use of Chlorohexidine for vaginal preparation surgery,

due to its labeling as a cause for irritation, studies have shown that when 2-4% Chlorhexidine is

used in the vaginal area there are little to no signs of irritation and the bacteria counts post

incision are less than the bacterial counts for povidone iodine<sub>1,2</sub>. Baby shampoo can also be used

as an effective antiseptic scrub with no irritation and no statistical difference in bacterial count

reduction as compared to povidone-iodine3. Little research has been done to look at the antiseptic

power of Chloroxylenol in vaginal surgeries. However, when used as a root canal antiseptic it

can reduce bacteria counts by 99.9%4. This is illustrative of its capability to reduce bacteria on a

mucus membrane similar to the vagina.

There is literature that shows the antiseptic power of Betadine, Peridex, Baby shampoo and

TechniCare for post-incisional bacteria counts, but little is known about the pre-incisional power

of these scrubs for vaginal access surgeries.

SPECIFIC AIMS OR OBJECTIVES

The aim of this study is to understand the power of vaginal surgical scrubs before and

after procedure completion. This will be done by collecting bacterial samples before antiseptic

preparation, 10 minutes after antiseptic preparation, and after completion of the procedure along

with follow-up data of irritation, infection post-surgery, and infection risk factors of each patient.

SIGNIFICANCE TO PATIENT, INSTITUTION, PROFESSION, OR ALL

Version: 6

Vaginal preparation research provides beneficial knowledge to hospitals and physicians in the prevention of surgical site infections (SSI). This specific project will provide insight regarding the bacteria-eliminating power of four different surgical scrubs used on the vaginal mucous membrane. There is potential for this study to determine the most effective scrub for vaginal surgeries, as well as correlate pre-procedure bacterial counts and likelihood of surgical site infections. The information collected from this study could benefit future patients and hospitals alike in terms of reducing the risk of SSI's. The risks of this study could be unidentified allergies to any of the surgical scrubs, or a loss of patient data. These are unlikely risks due to the protocol of the study.

## **METHODS**

This study will use block randomization. There will be four arms of the study one for each of the four surgical scrubs. There will be approximately 15 patients per arm. Patients undergoing surgeries which require a vaginal antiseptic preparation will be recruited from Wright State Physicians Obstetrics and Gynecology as well as other participating groups at Miami Valley Hospital. Procedures included in the study are procedures in which a vaginal preparation is performed, including procedures with a vaginal incision (hysterectomy, incontinence procedures), as well as general laparoscopic procedures (diagnostic laparoscopy, salpingectomy, oophorectomy, etc). Procedures excluded from the study are procedures which involve: any local infectious process such as cellulitis or abscess, have significant risk of washout of the vaginal preparation (hysteroscopy or vaginoscopy), any procedures for invasive cancer diagnoses, or procedures with significant risk of bleeding such as dilation and curettage (both for sampling or pregnancy-related), or endometrial ablation. Revision surgeries will also be excluded to decrease any complications. Patients who consent to the study will be given a ID and

Version: 6

will be randomly assigned to one of the four arms. Patients will be excluded if an allergy to any of the scrubs is listed or found. Each recruited patient will be over the age of 18 with ability to consent on their own.

Each patient will be given a standard prophylaxis 30 minutes before surgery. After prophylaxis administration and before surgical antiseptic preparation, a 10 second swab will be taken of the vagina making sure to span the surface area of the vaginal canal with avoidance of the cervix. The swab will then be broken off into a tube labeled with the patient ID, date, and "pre-scrub." The patient will then undergo antiseptic preparation with the assigned surgical prep. A standard procedure of application will be done for each of the arms. Ten minutes after application, another swab will be taken using the same procedure as the "pre-scrub" swab. This swab will be broken off in a tube labeled with the patient ID, date, and "post-scrub." Following the conclusion of the procedure, a third swab will be taken using the same procedure as the two pre-incision swabs. The third swab will then be broken off into a tube labeled with the patient ID, date, and "post-procedure-swab." The swabs will then be transported to CompuNet where they will be analyzed for aerobic, anaerobic bacteria and fungal colonies using Matrix Assisted Depolarization/Ionization Time of Flight mass spectrometry (MALDI-TOF).

The data of colony counts will be collected from CompuNet. BMI, age, prophylaxis, postmenopausal information, diabetic information, smoking history, surgical duration, complication in surgery, and length of hospital stay will all be collected from patient records. No patient identifiers will be collected<sub>5</sub>. Patients will be followed up on their surgery approximately two days, two weeks and a month after surgery to get information on irritation and/or surgical infection. This data will be collected either be phone call or at post-surgical follow-up appointment at Wright State Physicians. The South Hampton Grading Scheme for Surgical

Version: 6

Wounds will be used to Quantify Each patients level of irritation and/or infection. The scale is a

Zero to Five score, with Zero being no irritation or infection and Five being severe irritation or

infection<sub>15</sub>.

One potential obstacle of this study could be recruitment of patients. Patients will not be

given incentive for participation and will not acquire any direct benefit from the study. Another

potential issue may arise from the size of the study; there may not be enough subjects recruited

for each arm of the study to find a detectable and significant difference in the use of one surgical

scrub over another. There may also not be sufficient power to detect a difference in the risk of

post-operative surgical site infections.

Precautions will need to be taken for allergies. A recruited patient may not be aware of

personal allergies to the surgical scrubs. This would put the patient in harm if they are assigned

to a scrub that they are allergic to. Since data will be collected from the patient's medical

records, precautions will be taken to avoid loss of patient identifiers. All research investigators

will only utilize the patients assigned research ID. This will both protect the patient and avoid

bias.

**Statistical Analysis Plan** 

Bacterial and fungal colony counts will be coded as positive if counts are ≥5000 colonies/mL

and negative if < 5000 colonies. Statistical analyses will be conducted as follows:

Baseline charasteristics will be compared with Chi square (categorical data) and ANOVA

(continuous data) to determine potential differences for demographic and clinical characteristics

and for colony counts (positive vs negative) at the pre-scrub sample collection.

Each of the 3 target scrubs (baby shampoo, chlorhexidine and chloroxynel) will be compared to

povidone-iodine as the standard of care using Fisher's Exact tests for each pair comparison at the

Version: 6

post-scrub and post-procedure collections.

## REFERENCES

 Culligan PJ, Kubik K, Murphy M, Blackwell L, Snyder J. A randomized trial that compared povidone iodine and chlorhexidine as antiseptics for vaginal hysterectomy. Am J Obstet Gynecol. 2005 Feb;192(2):422-5.

2. Al-Niaimi A, Rice LW, Shitanshu U, Garvens B, Fitzgerald M, Zerbel S, et al. Safety and tolerability of chlorhexidine gluconate (2%) as a vaginal operative preparation in patients undergoing gynecologic surgery. Am J Infect Control. 2016 Sep 1;44(9):996-8.

 Garcia GA, Nguyen CV, Yonkers MA, Tao JP. Baby shampoo versus povidone-iodine or isopropyl alcohol in reducing eyelid skin bacterial load. Ophthal Plast Reconstr Surg.
 2017 Jan 6.

4. Lewis LA, Lathi RB, Crochet P, Nezhat C. Preoperative vaginal preparation with baby shampoo compared with povidone-iodine before gynecologic procedures. J Minim Invasive Gynecol. 2007 Nov-Dec;14(6):736-9.

- 5. Schafer E, Bossmann K. Antimicrobial efficacy of chloroxylenol and chlorhexidine in the treatment of infected root canals. Am J Dent. 2001 Aug;14(4):233-7.
- American College of Obstetricians and Gynecologists Women's Health Care Physicians,
   Committee on Gynecologic Practice. Committee opinion no. 571: Solutions for surgical preparation of the vagina. Obstet Gynecol. 2013 Sep;122(3):718-20.
- 7. Van Wicklin SA. Preoperative vaginal preps with chlorhexidine gluconate solution.

  American Journal of Obstetrics and Gynecology 2006 August 2006;195(2):624.

Version: 6

- 8. Vorherr H, Ulrich JA, Messer RH, Hurwitz EB. Antimicrobial effect of chlorhexidine on bacteria of groin, perineum and vagina. J Reprod Med. 1980 Apr;24(4):153-7.
- 9. Culligan P, Heit M, Blackwell L, Murphy M, Graham CA, Snyder J. Bacterial colony counts during vaginal surgery. Infect Dis Obstet Gynecol. 2003;11(3):161-5.
- 10. ALY R, MAIBACH H. Comparative antibacterial efficacy of a 2-minute surgical scrub with chlorhexidine gluconate, povidone-iodine, and chloroxylenol sponge-brushes. Am J Infect Control. 1988 AUG;16(4):173-7.
- 11. Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. national nosocomial infections surveillance system. Am J Med. 1991 Sep 16;91(3B):152S-7S.
- 12. Faro C, Faro S. Postoperative pelvic infections. Infect Dis Clin North Am. 2008 Dec;22(4):653,63, vi.
- 13. Kjolhede P, Halili S, Lofgren M. Vaginal cleansing and postoperative infectious morbidity in vaginal hysterectomy. A register study from the swedish national register for gynecological surgery. Acta Obstet Gynecol Scand. 2011 Jan;90(1):63-71.
- 14. Steiner HL, Strand EA. Surgical-site infection in gynecologic surgery: Pathophysiology and prevention. Obstet Gynecol. 2017 AUG;217(2):121-8.
- 15. Bailey IS, Karran SE, et al. Community surveillance of complications after hernia surgery. BMJ. 1992; 304: 469-471. (Table I, page 470)

Version: 6